CLINICAL TRIAL: NCT02486731
Title: Consequences of Noonan Syndrome/LEOPARD Syndrome Associated Shp2 Mutations on Different Signaling Pathways Activation: Relationship With Hormonal Sensitivity
Brief Title: Hormonal Sensitivity in Patients With Noonan and LEOPARD Syndromes
Acronym: NOLEO
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C13-59; 2013-A01428-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-03-04; First posted 2015-07-01 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Noonan Syndrome; LEOPARD Syndrome
Keywords: Hormonal sensitivity; bone growth
MeSH Terms: conditions — Noonan Syndrome; LEOPARD Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fibroblasts, adipocytes, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Noonan syndrome: Patients with Noonan syndrome
- LEOPARD syndrome: Patients with LEOPARD syndromes
- Controls: Healthy subjects

SUMMARY:
Noonan and LEOPARD syndromes share, with variable severity, different clinical traits, notably craniofacial manifestations, cardiopathies, short stature, and juvenile cancers.

The main genetic cause of these syndromes is missense mutation of the gene encoding the ubiquitous tyrosine phosphatase Shp2, found in more than half the patients with NS and in 80% of LS cases. Shp2 plays pivotal roles in development, growth, and metabolism by regulating key signalling pathways (Ras/Mitogen activated protein kinase (MAPK), Phosphoinositide-3 Kinases (PI3K)/Akt) in response to growth factors/hormones. Deregulation of these signalling pathways has been causally linked to NS and LS pathophysiology.

This project aims at better understanding hormonal sensitivity abnormalities in patients with Noonan syndrome (NS) or LEOPARD syndrome (LS) caused by mutations of the tyrosine phosphatase Shp2.

To reach this goal, the investigators will take advantage of different tissues (fibroblasts ± adipocytes) from patients with NS / LS compared to healthy controls.

All patients will have a skin biopsy and only patients about to undergo surgery will have a adipose tissue biopsy.

DETAILED DESCRIPTION:
The activation of different signaling pathways (Ras/MAPK, PI3K/Akt) in response to growth factors/hormones (growth hormone, insulin) in fibroblasts and/or in adipocytes from patients with NS or LS will be compared to those of healthy subjects.

These data will be correlated to clinical, hormonal, and biochemical characteristics of patients

ELIGIBILITY:
Inclusion Criteria:

Patients with Noonan syndrome (NS) or LEOPARD syndrome (LS):

* female or male
* age between 5 to 15 years
* clinical diagnosis of NS or LS according to published criteria
* signed informed consent of parents

Healthy controls:

* female or male
* age between 5 to 15 years
* no personal history of syndrome or chronic disease
* planned surgical procedure
* signed informed consent of parents

Exclusion Criteria:

* age below 5 or above 15 years
* pregnancy

In healthy controls: syndromic or chronic disease

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Data collected in patients with Noonan or LEOPARD syndromes will be compared to data of healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Phosphorylation of Erk and Akt in fibroblasts | Baseline
  To evaluate different signaling pathways activation (Ras/MAPK, PI3K/Akt) in response to growth factors/hormones (growth hormone, insulin) in fibroblasts from patients with NS or LS compared to healthy controls

SECONDARY OUTCOMES:
Phosphorylation of Erk and Akt in adipocytes | Baseline
  To evaluate different signaling pathways activation (Ras/MAPK, PI3K/Akt) in response to growth factors/hormones (growth hormone, insulin) in adipocytes from patients with NS or LS compared to healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- CIC de Toulouse- Unité pediatrique, Toulouse, France